CLINICAL TRIAL: NCT05467345
Title: Evaluation of the Performance of CONTOUR NEXT® and CONTOUR PLUS ELITE® Blood Glucose Monitoring Systems (BGMS) in Neonates Using Capillary Blood Samples
Brief Title: Evaluation of the Performance of CONTOUR NEXT® and CONTOUR PLUS ELITE® BGMS in Neonates Using Capillary Blood Samples
Status: Completed | Type: Observational
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: GCA-PRO-2021-003-01
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Contour Next and Contour Plus Elite BGMS testing of neonatal blood — The purpose of this study is to extend the intended use of two BGMSs to include testing of neonatal blood by Health Care Professionals in a clinical setting for the quantitative measurement of glucose levels in neonates.

SUMMARY:
The purpose of this study is to extend the intended use of two BGMSs to include testing of neonatal blood by Health Care Professionals in a clinical setting for the quantitative measurement of glucose levels in neonates.

DETAILED DESCRIPTION:
This trial will evaluate the performance of both the CONTOUR NEXT BGMS and CONTOUR PLUS ELITE BGMS using blood from neonates within a hospital ward, e.g. routine/newborn nurseries, Special Care Nurseries, Neonatal Intensive Care Unit (NICU). The investigational BGMSs will be tested by a Point-of-Care operator using residual heel-stick capillary blood samples from neonates who underwent routine prescribed testing.

ELIGIBILITY:
Inclusion Criteria:

* Residual capillary (heel-stick) blood samples from neonates (less than 28 days of age) after birth as part of prescribed testing.
* Sample blood volume must be sufficient to complete investigational testing in addition to routine prescribed clinical laboratory testing.

Exclusion Criteria:

* Samples from subjects who are ≥ 28 days of age.
* Samples from subjects who have previously been enrolled into this study.

Ages: 0 Days to 27 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The subject population will consist of neonates from hospital wards (e.g. routine/newborn nurseries, SCN, NICU) of the clinical investigational site.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Dietzen, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, Washington University, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: blood samples
Groups:
- Testing of Neonatal Blood With BGMS: The neonatal blood will be tested on two different BGMS: 1) Contour Next BGMS and 2) Contour Plus Elite BGMS. Each blood sample will be tested in duplicate on each BGMS. The results will be compared to the laboratory reference result.
Period: Overall Study
Arm/Group | Testing of Neonatal Blood With BGMS
Started | 120; 240 blood samples
Completed | 120; 240 blood samples
Not Completed | 0; 0 blood samples

BASELINE CHARACTERISTICS:
Population: 120 participants were enrolled in the study. Each participant provided 2 blood samples that were tested. So, the number of results analyzed is 240.
Units Other Than Participants: blood samples
Groups:
- Testing of Neonatal Blood With BGMS: The neonatal blood will be tested on two different BGMS: 1) Contour Next BGMS and 2) Contour Plus Elite BGMS. The results will be compared to the laboratory reference result.
Arm/Group | Testing of Neonatal Blood With BGMS
Number analyzed (Participants) | 120
Number analyzed (blood samples) | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 120
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 67
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Results From the Contour Next BGMSs Reference Values Within ±12.5% of Reference Values
Description: At least 95% of all blood glucose results shall fall within ±12.5% of reference values (laboratory method) for glucose concentration ≥100 mg/dL(5.55 mmol/L )and within ±12 mg/dL(±0.67 mmol/L) at glucose concentrations <100 mg/dL(5.55 mmol/L).
Time Frame: 1 day
Population: Neonates in a hospital neonatal unit.
Measure: Count of Units; unit: blood samples
Units Other Than Participants: blood samples
Arm/Group | Testing of Neonatal Blood With BGMS
Number analyzed (Participants) | 120
Number analyzed (blood samples) | 240
blood samples | 240

2. Primary Outcome: Number of Results From the Contour Plus Elite BGMSs Reference Values Within ±12.5% of Reference Values
Description: At least 95% of values should be within ±12.5% of reference values (laboratory method) for glucose concentration ≥75 mg/dL(4.16 mmol/L) and within ±15 mg/dL(±0.83 mmol/L) at glucose concentrations < 75 mg/dL(4.16 mmol/L).
Time Frame: 1 day
Population: Neonates in a neonatal hospital ward.
Measure: Count of Units; unit: blood samples
Units Other Than Participants: blood samples
Arm/Group | Testing of Neonatal Blood With BGMS
Number analyzed (Participants) | 120
Number analyzed (blood samples) | 240
blood samples | 240

ADVERSE EVENTS:
Time Frame: 1 day
Description: No adverse reactions expected since the samples were leftover blood. No contact with the neonate was made.
Arm/Group | Testing of Neonatal Blood With BGMS
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT05467345/Prot_SAP_000.pdf